CLINICAL TRIAL: NCT07057154
Title: Glycatetd Hemoglobin Index and Red Cell Distribution Width as Prognstic Indicator in Critical Ill Patients
Brief Title: Glycated Hbg Index and RDW as Prognstic Indicator in Critical Ill Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rania Moukhter aziz aldean, Doctor, Assiut University
Other Study IDs: Rule of HBGA1C in critical ill
Record Dates: First submitted 2025-05-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Critical Ill Patients
MeSH Terms: interventions — Erythrocyte Indices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hbg and RDW — Hbg and RDW as prognstic indicator in critical ill patients

SUMMARY:
The aim of this study was to evaluate the impact of GHI and RDW as prognostic indicator in critically ill Patients.

DETAILED DESCRIPTION:
Primary (Main): determine the levels of the GHI And RDW In Critically Ill Patients at Critical and intermediate care units.

b. Secondary (Subsidiary): Evaluate the prognostic significance of these parameters on patient outcomes, such as overall survival, progression-free survival, response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. patients admitted to Critical and Intermediate Care Units in Internal Medicine Department after history taking, examination and diagnosis
2. diabtic Patients 3-animic Patients

Exclusion Criteria:

* Patients under 18 years of age
* ICU stay < 24 h
* patients without HbA1c, FBG, or RDW data or anything's that's affect the HbA1c .

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients except patients in exculcion critira
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2025-07-05 (Estimated); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Glycated Hemoglobin level | Baseline
  Measurement of Hb level in all patients upon ICU admission.
Red Cell Distribution Width (RDW) | baseline
  Measurement of RDW in all patients upon ICU admission.
Hemoglobin (Hb) Level | baseline
  Measurement of Hb level in all patients upon ICU admission.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — https://zumj.journals.ekb.eg/article_322723_e4dc2f307e76021f9d66ea9214c322a1.pdf
- See also: Related Info — https://www.njmonline.nl/getpdf.php?id=1376